CLINICAL TRIAL: NCT06332222
Title: Recovery With Tart Cherry Supplementation Following a Marathon.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Iprona Lana SpA (Unknown)
Responsible Party: Principal Investigator, Glyn Howatson, Professor Glyn Howatson, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1987
Record Dates: First submitted 2024-03-11; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Exercise Recovery
Keywords: Muscle Damage; Inflammation; Tart Cherry; Intervention; Marathon
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vistula Tart Cherry (Active Comparator): Supplemented with tart cherries.
  Interventions: Dietary Supplement: Tart Cherry
- Placebo (Placebo Comparator): Supplemented with a calorie matched placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Tart Cherry — 7 day supplementation
  Arms: Vistula Tart Cherry
Other: Placebo — 7 day supplementation
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare recovery in healthy, active runners.

The main questions it aimed to answer were whether 7 day supplementation with Vistula TC attenuated:

* muscle function
* inflammation
* soreness following a marathon run.

Participants will either consume a spray-dried tart cherry supplement or a calorie-matched placebo-control for 7 days, and complete a marathon. Participants will perform functional tests, be assessed for their perceptual recovery and markers of inflammation and muscle damage via:

* maximal voluntary contractions
* counter movement jumps
* visual analog scales to assess soreness
* blood samples

DETAILED DESCRIPTION:
Participants

Participants were recruited from a pool of runners taking part in the Kielder marathon, Northumberland, UK. Based on a previous study that examined the effects of TC on recovery after a marathon race, it was estimated that at 0.80 power and 0.05 significance, the minimum number of participants required to detect a ≥10% group difference (SD 8%) in one of our primary outcomes, MVC, would be n = 13 per group. Thirty-eight participants were initially recruited and provided written, informed consent. Three withdrew after baseline assessment, two due to illness and one that did not want to use the intervention before the race. Therefore, 35 recreationally active runners took part in this double-blind, randomized, placebo-controlled, independent group design study. The participants were asked to maintain their habitual diet, and to fill in a short food log when they consumed foods/drinks, that were typically high in polyphenols, such as fruits & vegetables, fruit juices, nuts and seeds, chocolate and coffee/tea. Participants were asked to refrain from strenuous exercise (other than completing training runs before the marathon) for the duration of the study and to refrain from non-steroidal anti-inflammatory or analgesic drugs, and nutritional such as protein, and vitamins. This study received ethical approval from Northumbria University Ethics Committee (reference number: 1987) and it was registered as a clinical trial with clinicaltrials.gov (TBC).

Experimental Design

The study design was an independent group design that was double blinded, randomized, and placebo controlled. Participants were assigned to two groups to consume either the TC capsules or a placebo capsule, matched for calorific content. Participants were required to attend the laboratory for a familiarisation, baseline assessment (which took place 5-6 days before the race), and 24- and 48-h post-marathon. Participants had an assessment of their functional and perceptual measures of recovery, pre-, immediately post-, 24- and 48- h post-marathon. The loading phase for the intervention ingestion commenced four days prior to the marathon and on the day of the marathon, as well as the two days following, totaling seven days.

Marathon Characteristics

The marathon took place at Kielder Water, Northumberland, UK on the 08/10/23, and consisted of an almost entirely off-road course around northern Europe's largest man-made lake, Kielder Water, with a total ascent of 613 m and total descent 616 m. The environmental conditions on the day of the race were: barometric pressure, 1023 mb; temperature, 16 C; wind speed, 7 km/h; humidity, 99%. The conditions were wet under foot and there was a mist in the air causing reduced visibility (50 m).

Treatment and Dietary Control

The participants consumed either a placebo or a TC spray-dried extract made from a variety of TC know as 'Nadwiślanka' also called Vistula Cherries (extract brand name CherryCraft®, Iprona Lana SpA, South Tyrol, Italy). The invention was consumed in the form of capsules, twice per day for a period of seven days. The supplementation period was similar to previous studies and are summarized in a recent meta-analysis. The dose increased on the day of the damaging stimuli to increase the bioavailability of phytochemicals when exercise stress and its repercussions were elevated; previous bioavailability studies have shown that increasing the dose can elevate anthocyanin and phenolic acids. The participants were required to consume a lower dose (73.5 mg of anthocyanins, according to manufacturers data) for the first four days, then consume a higher dose (132.3 mg of anthocyanins, according to manufacturers data) for the remaining three days (day of marathon protocol, 24 and 48 h post). The loading dose was determined by replicating the average reported anthocyanin content from previous studies which used powdered TC products , which was 77 mg. Then the higher dose was approximately double, similarly to the papers which have observed some differences in dose-response relationship studies.

Functional Performance and Perceptual Variables

After a familiarisation (one week prior to baseline assessments), participants were assessed for their fatigue and recovery via measures of functional performance and perceptual variables at baseline (5-6 days prior to the race), immediately post, 24- and 48-h post- marathon.

Maximal Voluntary Contraction (MVC)

MVC was measured with a portable strain gauge (MIE Medical Research Ltd., Leeds, UK). All assessments were performed with the participants seated in an upright position. After adjusting the strap to ensure a 90° knee joint angle was attained (verified with a goniometer), participants were instructed to push against the strap with maximal force for a 3 s contraction. The peak value (N) from three maximal contractions (separated by 30 s) was used for analysis. Verbal encouragement was provided for all assessments.

Counter Movement Jump (CMJ)

CMJ height was measured using an Optojump system (Microgate, Bolzano, Italy), which calculated jump height (cm) via flight time. When performing the jumps, participants were instructed to keep their hands on their hips throughout the full movement. Participants were required to descend into a squat and jump vertically with maximum effort. Three maximal efforts were performed, separated by 30 s of passive (standing) recovery, and the average value was used for data analysis.

Active Muscle Soreness

Delayed onset muscle soreness (DOMS) of the participants lower limbs was assessed via the use of a 200 mm visual analogue scale (VAS). Participants rated their lower limb soreness after performing one squat (at approximately 90° knee flexion) on a line with the far-left end point representing 'no pain' (0 mm) and the far-right end point representing 'extremely painful' (200 mm).

Passive Perceptual Wellness Variables

While seated the participants rated their feelings of soreness (passive), fatigue, energy sleepiness and readiness to train using a VAS with the far-left end point representing 'not at all' (0 mm) and the far-right end point representing 'extremely' (200 mm).

Blood Sampling Procedure

Venous blood samples were collected from a vein at antecubital fossa on four occasions (pre, immediately post, 24 and 48 h post the marathon). Samples were immediately centrifuged (3000 × g rpm) at 4°C for 15 min and the supernatant was aspirated into aliquots and then stored at -80°C until analysis. Serum was later analysed for CK and hs-CRP using an automated device (Cobas c702, Roche Diagnostics, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Active

Exclusion Criteria:

* Food allergy
* Smokers
* Cardiovascular/gastrointestinal/thyroid/renal disease
* Musculoskeletal injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Contraction | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Leg extension MVC to measure functional recovery

SECONDARY OUTCOMES:
Counter Movement Jump | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Jump height assessment to measure functional recovery
Active Muscle Soreness | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Visual analog scale to assess perceptual soreness, on a standard 200 mm line with the far-left end point representing 'no pain' (0 mm) and the far-right end point representing 'extremely painful' (200 mm).
Serum Concentration of High-Sensitive C-Reactive Protein | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Blood sample to measure inflammation
Serum Concentration of Creatine Kinase | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Blood sample to measure indirect muscle damage
Perceptual Measures | Measurements were taken on 4 separate occasions. Once at baseline, before supplementation began, which took place 5-6 days before the race. The measurement was taken again immediately post the marathon and again 24 and 48 hours post marathon.
  Assessed via visual analog scales: soreness (passive), fatigue, energy sleepiness and readiness to train. Using a standard 200 mm line, participants rated the aforementioned perceptions, with the far-left end point representing 'not at all' (0 mm) and the far-right end point representing 'extremely' (200 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levers K, Dalton R, Galvan E, O'Connor A, Goodenough C, Simbo S, Mertens-Talcott SU, Rasmussen C, Greenwood M, Riechman S, Crouse S, Kreider RB. Effects of powdered Montmorency tart cherry supplementation on acute endurance exercise performance in aerobically trained individuals. J Int Soc Sports Nutr. 2016 May 26;13:22. doi: 10.1186/s12970-016-0133-z. eCollection 2016. PMID 27231439
- [Background] Howatson G, McHugh MP, Hill JA, Brouner J, Jewell AP, van Someren KA, Shave RE, Howatson SA. Influence of tart cherry juice on indices of recovery following marathon running. Scand J Med Sci Sports. 2010 Dec;20(6):843-52. doi: 10.1111/j.1600-0838.2009.01005.x. PMID 19883392
- [Background] Hill JA, Keane KM, Quinlan R, Howatson G. Tart Cherry Supplementation and Recovery From Strenuous Exercise: A Systematic Review and Meta-Analysis. Int J Sport Nutr Exerc Metab. 2021 Mar 1;31(2):154-167. doi: 10.1123/ijsnem.2020-0145. Epub 2021 Jan 13. PMID 33440334
- [Background] Hooper DR, Orange T, Gruber MT, Darakjian AA, Conway KL, Hausenblas HA. Broad Spectrum Polyphenol Supplementation from Tart Cherry Extract on Markers of Recovery from Intense Resistance Exercise. J Int Soc Sports Nutr. 2021 Jun 14;18(1):47. doi: 10.1186/s12970-021-00449-x. PMID 34126996
- [Background] Morehen JC, Clarke J, Batsford J, Barrow S, Brown AD, Stewart CE, Morton JP, Close GL. Montmorency tart cherry juice does not reduce markers of muscle soreness, function and inflammation following professional male rugby League match-play. Eur J Sport Sci. 2021 Jul;21(7):1003-1012. doi: 10.1080/17461391.2020.1797181. Epub 2020 Aug 6. PMID 32672095
- [Background] Wangdi JT, O'Leary MF, Kelly VG, Jackman SR, Tang JCY, Dutton J, Bowtell JL. Tart Cherry Supplement Enhances Skeletal Muscle Glutathione Peroxidase Expression and Functional Recovery after Muscle Damage. Med Sci Sports Exerc. 2022 Apr 1;54(4):609-621. doi: 10.1249/MSS.0000000000002827. PMID 34772901
- [Background] McCormick R, Peeling P, Binnie M, Dawson B, Sim M. Effect of tart cherry juice on recovery and next day performance in well-trained Water Polo players. J Int Soc Sports Nutr. 2016 Nov 14;13:41. doi: 10.1186/s12970-016-0151-x. eCollection 2016. PMID 27895542
- [Background] Kupusarevic J, McShane K, Clifford T. Cherry Gel Supplementation Does Not Attenuate Subjective Muscle Soreness or Alter Wellbeing Following a Match in a Team of Professional Rugby Union players: A Pilot Study. Sports (Basel). 2019 Apr 5;7(4):84. doi: 10.3390/sports7040084. PMID 30959854
- [Background] Abbott W, Brashill C, Brett A, Clifford T. Tart Cherry Juice: No Effect on Muscle Function Loss or Muscle Soreness in Professional Soccer Players After a Match. Int J Sports Physiol Perform. 2020 Feb 1;15(2):249-254. doi: 10.1123/ijspp.2019-0221. Epub 2019 Oct 28. PMID 31188696
- [Background] Bell, P. G., Gaze, D. C., Davison, G. W., George, T. W., Scotter, M. J., & Howatson, G. (2014). Montmorency tart cherry (Prunus cerasus L.) concentrate lowers uric acid, independent of plasma cyanidin-3-O-glucosiderutinoside. journal of functional foods, 11, 82-90. doi:10.1016/j.jff.2014.09.004
- [Background] Keane KM, Bell PG, Lodge JK, Constantinou CL, Jenkinson SE, Bass R, Howatson G. Phytochemical uptake following human consumption of Montmorency tart cherry (L. Prunus cerasus) and influence of phenolic acids on vascular smooth muscle cells in vitro. Eur J Nutr. 2016 Jun;55(4):1695-705. doi: 10.1007/s00394-015-0988-9. Epub 2015 Jul 11. PMID 26163338
- [Background] Levers K, Dalton R, Galvan E, Goodenough C, O'Connor A, Simbo S, Barringer N, Mertens-Talcott SU, Rasmussen C, Greenwood M, Riechman S, Crouse S, Kreider RB. Effects of powdered Montmorency tart cherry supplementation on an acute bout of intense lower body strength exercise in resistance trained males. J Int Soc Sports Nutr. 2015 Nov 16;12:41. doi: 10.1186/s12970-015-0102-y. eCollection 2015. PMID 26578852
- [Background] Kastello, G., Bretl, M., Clark, E., Delvaux, C., Hoeppner, J., McNea, L., & Strauss, J. (2014). The effect of cherry supplementation on Exercise induced oxidative stress. International Journal of Food Sciences and Nutrition, 1(1), 20-26.
- [Background] Clifford T, Bell O, West DJ, Howatson G, Stevenson EJ. Antioxidant-rich beetroot juice does not adversely affect acute neuromuscular adaptation following eccentric exercise. J Sports Sci. 2017 Apr;35(8):812-819. doi: 10.1080/02640414.2016.1192670. Epub 2016 Jun 7. PMID 27267689